CLINICAL TRIAL: NCT01603511
Title: Effectiveness of Heat Donation Through the Head or Torso on Mild Hypothermic Rewarming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr.Gordon Giesbrecht, Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2012:024; NSERC PIN (Other Grant/Funding Number: NSERC PIN)
Record Dates: First submitted 2012-05-18; First posted 2012-05-23 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Rewarming by Shivering Heat Production Only; Rewarming by External Heat to the Torso; Rewarming by External Heat to the Head
Keywords: rewarming; core cooling; afterdrop; pre-hospital treatment; hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Rewarming modality — A commercial charcoal heater will be applied to the torso or the head in two of the trials. The control trial involves shivering only.
  Other Names: Charcoal heater; STK Heatpac

SUMMARY:
The study will compare the rewarming effectiveness of heat donation through the head or the torso during rewarming of mildly hypothermic subjects. Warming will be accomplished through either forced-air warming or using a charcoal heater; both units are commonly used for warming. The investigators hypothesize that head warming will be as, or more, effective compared to

DETAILED DESCRIPTION:
Dr. Gordon Giesbrecht is studying/comparing the effectiveness of heat donation through the head or the torso in rewarming a mildly hypothermic individual. A rigid forced-air warming cover for the head or the torso will be used to rewarm the hypothermic individuals.

Subjects will be asked to participate in three experimental trials, separated by at least 48 hours. Each trial will last about 4 hours (1 hour for setup, 1 hour for cooling, and 2 hours for rewarming and removal of instrumentation).

On each of the three trials, subjects will undergo immersion to the level of the sternal notch in a tank of 8˚C water for up to 60 minutes. They will then exit the water, be dried off and lie in a hooded sleeping bag with the head inside the hood where one of the three warming procedures will be administered for 60 minutes or until core temperature returns to normal values ( ̴ 36.5-37˚C).

A. Spontaneous rewarming (Shivering Only) - In this control condition, no external heat will be provided and you will rewarm spontaneously with the heat produced from shivering.

B. Head Warming (Head): Either of these rewarming methods will be used:

* Forced-Air Warming to the Head (FAW-H) - A modified rigid forced-air warming cover will be placed over your head. Warm air ( ̴43˚C) will blow into the cover through an inlet on top of the cover and will escape from the bottom of the cover. You will be breathing warm air (̴ 43˚C).
* Charcoal Heater to the Head (CH-H) - A charcoal heater will be placed on right side of your face/head with ducts wrapping around the dorsum of the head, anteriorly over the forehead, nose, chin and the neck, not covering the eyes or the mouth. You will be breathing ambient air (̴ 22˚C).

C. Torso Warming - Either of these rewarming methods will be used:

* Forced-Air Warming to the Torso (FAW-T) - A specially designed portable rigid forced-air cover (PORIFAC) will be placed over your torso and the upper thighs. Warm air (̴ 43˚C) will blow into the cover through an inlet above the abdomen and will escape from the bottom of the cover. Participant will be breathing ambient air (̴ 22˚C).
* Charcoal Heater to the Torso (CH-T) - The charcoal heater will be placed on your anterior chest with a towel in between. The flexible ducts will be applied to the areas of high heat transfer i.e. over the shoulders, neck, and then anteriorly under the axillae to cross over the lower anterior chest. You will be breathing ambient air at room temperature (~22˚C).

After 60 minutes of warming, subjects will be placed in a warm water bath (40-42˚C) until they are comfortable and core temperature returns to normal values (̴ 36.5-37˚C).

Outcome measures include rate of core cooling, afterdrop amount, rate of rewarming, skin heat flux, oxygen consumption and shivering intensity.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 yrs old, males or females, healthy

Exclusion Criteria:

* cardiopulmonary disease
* any symptoms caused by cold exposure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Rate of body core rewarming | 60 minutes
  Esophageal temperature will be used to determine the rate of core temperature rewarming during 60 minutes of rewarming via either shivering only, or external heat donated to the torso or the head.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon G Giesbrecht, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada